CLINICAL TRIAL: NCT04390061
Title: TOFAcitinib Plus Hydroxycloroquine vs Hydroxycloroquine in Patients With Early Onset SARS-CoV2 (COVID-19) Interstitial Pneumonia:a Multicenter Randomized Controlled Open Label Trial
Brief Title: TOFAcitinib Plus Hydroxycloroquine vs Hydroxycloroquine in Patients With COVID-19 Interstitial Pneumonia
Acronym: TOFACoV-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Università Politecnica delle Marche (Other)
Collaborators: Azienda Ospedaliera Ospedali Riuniti Marche Nord (Unknown); Ospedale Civile Santo Spirito, Pescara (Unknown); Università Magna Grecia, Catanzaro (Unknown); ASST Papa Giovanni XXIII, Bergamo (Unknown); Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma (Unknown); ASST Cremona, Cremona (Unknown); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other); Ospedale di Circolo e Fondazione Macchi, Varese (Unknown)
Responsible Party: Principal Investigator, Armando Gabrielli, Full Professor Internal Medicine, Università Politecnica delle Marche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-002035-30
Record Dates: First submitted 2020-05-13; First posted 2020-05-15 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Pneumonitis, Interstitial; COVID-19
MeSH Terms: conditions — Lung Diseases, Interstitial; COVID-19 | interventions — tofacitinib; Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Multicenter open label randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tofacitinib+HYQ (Experimental): Tofacitinib 10mg cp twice a day + Hydroxychloroquine 200mg cp three times a day, both for 14 days
  Interventions: Drug: Tofacitinib; Drug: Hydroxychloroquine
- Hydroxychloroquine (Active Comparator): Hydroxychloroquine 200mg cp three times a day for 14 days
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Tofacitinib — Jak-1/3 inhibitor
  Other Names: Xeljanz
  Arms: tofacitinib+HYQ
Drug: Hydroxychloroquine — Standard Therapy

SUMMARY:
Multifocal interstitial pneumonia represents the most common cause of admission in intensive care units and death in SARS-CoV2 infections. In our Hospital, similarly to what reported in literature, up to 25% of admitted patients with pneumonitis requires mechanical ventilation or oro-tracheal intubation within 5-10 days. No established treatment is available for this condition. Preliminary evidence is accumulating about the efficacy of an aggressive treatment of the corona virus-induced inflammation and, in particular, investigators believe that blocking JAK1 is clinically rewarding in down-regulating IL-6 driven inflammation in patients with corona-virus infection. Thus, investigators designed a randomized controlled trial to test the hypothesis that adding Tofacitinib to the standard treatment in the early phase of COVID related pneumonitis could prevent the development of severe respiratory failure needing mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV2 Infection diagnosed by rt-PCR
* CT-scan confirmed interstitial pneumonia
* Hospital admission from less than 24h
* P/F ratio >150 mmHg
* Written Informed Consent

Exclusion Criteria:

* Age <18 ys or >65
* Patients in mechanical ventilation at time of admission
* Severe Hearth failure (NYHA 3 or 4)
* QTc > 470 ms or >500 ms in wide QRS patients
* Severe History of Chronic Ischemic Heart Disease, defined as history of Major Adverse Cardiovascular Event and/or recent (one year) revascularization.
* History of recurrent Deep Venous Thrombosis and Pulmonary Embolism or established thrombophilic conditions (e.g. history of anti-phospholipid antibodies, …)
* Active Bacterial or Fungal Infection
* Hematological cancer
* Metastatic or intractable cancer
* Pre-existent neurodegenerative disease
* Severe Hepatic Impairment,
* History of acute diverticular disease or intestinal perforation
* HBsAg positive and/or HBV-DNA positive patients
* Severe Renal Failure (Creatinine Clearance <30ml/h)
* Active Herpes zoster infection
* Patients with active or latent TB
* Severe anemia (Hb<9g/dl)
* Lymphocyte count below 750/mcl
* Neutrophil count below 1000/mcl
* Platelet count below 50000/mcl
* Pregnancy or Lactation
* History of intolerance to the experimental drugs or excipients
* Degenerative maculopathy or other relevant retinal disease
* Inability to give informed consent (severe transitory or permanent mental impairment, incapacitation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Prevention of severe Respiratory Failure requiring mechanical ventilation | 14 days
  Rate of patients needing mechanical ventilation to maintain PaO2/FIO2>150

SECONDARY OUTCOMES:
Prevention of need of ICU admission | 28 days
  Rate of patients needing admission to the intensive care unit
Prevention of COVID-19 related Deaths | 28 days
  Rate of patients who die due to COVID-19 related conditions
Identification of predictors of outcome | 14 days
  Role of some clinical and laboratory factors in predicting outcome (Age, sex, smoking status, Body Mass Index (BMI), Comorbidities (Diabetes, number of comorbidities), Respiratory Failure at admission defined as PaO2/FiO2<300, Extension of Ct-scan involvement, basal level of serum IL-6, vW-Factor, Thrombomodulin, KL-6, sACE2 and SP-D )
Incidence of Treatment-Emergent Adverse Events | 28 days
  Rate of severe drug-related adverse events

IPD SHARING:
Plan to Share IPD: No